CLINICAL TRIAL: NCT03361852
Title: A Pilot Study of a Personalized Neoantigen Cancer Vaccine in Combination With Pembrolizumab Following Front-Line Rituximab in Follicular Lymphoma
Brief Title: Personalized Neoantigen Cancer Vaccine + Pembrolizumab After Rituximab for Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Reid Merryman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-353
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: All patients will receive 4 weekly doses of rituximab. Afterwards, will receive either NeoVax alone (first 5 patients) or NeoVax in combination with pembrolizumab (5 patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neo Vax (Experimental): * Neo Vax is injected into up to 4 different anatomic site.
  * NeoVax may be administered within +/- 1 day of the scheduled administration date for days 4 and 8,
  * Within +/-3 days of the scheduled administration date for days 15 and 22
  * Within +/-7 days of days 78 and 134.
  * Participants will receive Rituximab weekly x 4 weeks per institutional standard
  Interventions: Drug: Rituximab; Biological: Neo Vax
- NeoVax and pembrolizumab (Experimental): * Neo Vax is injected into up to 4 different anatomic site.
  * NeoVax may be administered within +/- 1 day of the scheduled administration date for days 4 and 8,
  * Within +/-3 days of the scheduled administration date for days 15 and 22
  * Within +/-7 days of days 78 and 134.
  * Patients will receive pembrolizumab every 3 weeks starting on day 78
  * Participants will receive Rituximab weekly x 4 weeks per institutional standard
  Interventions: Drug: Rituximab; Biological: Neo Vax; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Rituximab — Rituximab is classified as a monoclonal antibody. It works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells
  Other Names: Rituxan
Biological: Neo Vax — Neo Vax is an experimental "viral mimic" and an activator of immunity.
Drug: Pembrolizumab — Pembrolizumab is a monoclonal antibody that targets PD-1. It is a type of immunotherapy
  Arms: NeoVax and pembrolizumab

SUMMARY:
This research study is studying a novel type of FL vaccine as a possible treatment for follicular lymphoma (FL).

The agents involved in this study are:

* Rituximab
* Personalized NeoAntigen vaccine
* Poly-ICLC
* Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining the Personalized Neoantigen Vaccine (NeoVax) in patients diagnosed with follicular lymphoma. The FDA (the U.S. Food and Drug Administration) has not approved the Personalized Neoantigen Vaccine as a treatment for any disease.

Patients will receive 4 weekly doses rituximab (a CD20 monoclonal antibody) during NeoVax manufacturing (see below). Patients who have stable disease or achieve a response with rituximab therapy will next receiving NeoVax alone (first 5 patients) or NeoVax in combination with pembrolizumab (a PD-1 monoclonal antibody).

The purpose of this study is to determine if it is possible to make and safely administer a vaccine against FL by using information gained from specific genetic characteristics of the participant's own FL cells. The investigators plan to analyze the specific genetic characteristics of the participant's own FL cells and use that information to produce proteins that may help the participant's immune system recognize and fight FL cells.

This vaccine has already been tested in clinical trials in patients with advanced melanoma (a type of skin cancer) and glioblastoma (a type of brain cancer). The current study will examine the ability of the vaccine to stimulate the participant's immune system when given at several different timepoints, and will examine the participant's blood cells for signs that the FL has changed or decreased.

FL cells will be obtained from a tumor biopsy. The genetic material contained in the FL cells will be examined for the presence of tumor-specific mutations. This information will be used to prepare small protein fragments, which are called "peptides." The vaccine will consist of up to 20 of these peptides as well as a drug called Poly-ICLC. A peptide from the tetanus vaccine will also be included to boost the immune response.

Poly-ICLC (also called Hiltonol) is an experimental "viral mimic" and an activator of immunity. Poly-ICLC binds proteins on the surface of certain immune cells to make it appear as if a virus is present. When the cells detect the vaccine, they think it is a virus and turn on the immune system. Poly-ICLC will be mixed with NeoAntigen peptides and administered as an injection given underneath the skin. Poly-ICLC is an investigational drug, meaning the FDA has not approved it as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade I-IIIA follicular lymphoma (pathology must be confirmed at DFCI/BWH)
* Planned treatment with 4 weekly doses of rituximab.
* No prior systemic therapy for follicular lymphoma; prior radiation with palliative or curative intent is allowed if radiation occurred more than 3 months prior to study entry
* Patient must have measurable disease by Cheson criteria
* Age ≥ 18 years.
* ECOG performance status < 2.
* Participants must have normal organ and marrow function as defined below:

  * Hemoglobin > 9 gm/dl (ESAs or transfusion are not allowed) [greater than 8 gm/dl if there is lymphoma involvement of the bone marrow]
  * ANC > 1000 (greater than 750 if there is lymphoma involvement of the bone marrow)
  * Platelet count >100,000 (greater than 50,000 if there is lymphoma involvement of the bone marrow]
  * International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) < 1.5 x ULN unless subject is on anticoagulation as long as PT or aPTT is within intended therapeutic range of anticoagulant used
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal (< 5 x ULN if there are hepatic metastases)
  * Creatinine < 1.5 x ULN or measured or calculated creatinine clearance (GFR can also be used in place of creatinine clearance) > 30 ml/min for subject with creatinine > 1.5 x institutional ULN
  * total bilirubin less than institutional 1.5 x ULN (or a direct bilirubin < ULN if total bilirubin is >1.5 x ULN)
* The effects of NeoVax and poly-ICLC on the developing human fetus are unknown. For this reason, women of childbearing potential (WOCBP) must have a negative pregnancy test (serum) before entry onto the trial and within 7 days prior to start of study vaccination.
* Female patients enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity throughout the study, starting with visit 1 through 4 weeks after the last dose of study therapy. Approved contraceptive methods include for example; intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception. Male participants need to agree to use an adequate method of contraception
* Patient is agreeable to allow tumor (from peripheral blood, lymph node, or effusion) and normal tissue (from saliva) samples to be submitted for complete exome and transcriptome sequencing.
* Ability to understand and the willingness to sign a written informed consent document.

Additional Inclusion Criteria for Treatment Registration

* Participants must meet the following criteria (in addition to the above) to be eligible to proceed to receive vaccine treatment on the study:
* At least 7 immunizing peptides can be designed
* Continue to meet inclusion and exclusion criteria for Screening Registration (note: hepatitis B and hepatitis C serologies do not need to be repeated unless there is a clinical concern that an exposure has occurred since the screening phase).
* Achieved a CR, PR, or SD with no residual mass greater than 5 cm per Lugano criteria following single agent rituximab per

Exclusion Criteria:

* Recovered from all AEs due to rituximab to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Prior systemic therapy for follicular lymphoma with the exception of 4 weekly doses of rituximab as proscribed per protocol
* Radiation with palliative or curative intent within 90 days of study screening
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Participants who are receiving any other investigational agents.
* Previous bone marrow or stem cell transplant
* Concomitant therapy with immunosuppressive or immunomodulatory agents; chronic use of systemic corticosteroids at doses of 10 mg of prednisone (or equivalent) for indications other than treatment of follicular lymphoma is acceptable. Use of higher doses of corticosteroids after initial registration is acceptable if tapered to 10 mg of prednisone (or equivalent) or les at least 7 days prior to NeoVax administration so long as the corticosteroids were not administered for follicular lymphoma.
* Use of a non-oncology vaccine therapy for prevention of infectious diseases within 2 weeks prior to any NeoVax administration.
* History of severe allergic reactions attributed to any vaccine therapy for the prevention of infectious diseases.
* Active, known, or suspected autoimmune disease or immunosuppressive conditions with the exception of vitiligo, type 1 diabetes, residual autoimmune-related hypothyroidism requiring hormone replacement, or psoriasis not requiring systemic treatment.
* Progressive disease or stable disease with residual tumor mass > 5 cm by CT scan (measured as long axis) following 4 weekly doses of rituximab (for treatment phase only).
* Any documented transformation to diffuse large B cell lymphoma or grade 3Bfollicular lymphoma.
* Currently requiring chronic intravenous immunoglobulin G (IVIG)
* Active infection with hepatitis B or C (see Study Calendar in Section 10 for screening assays).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* Any underlying medical condition, psychiatric condition or social situation that in the opinion of the investigator would compromise study administration as per protocol or compromise the assessment of AEs.
* Pregnant women are excluded from this study because personalized neoantigen peptides and poly-ICLC are agents with unknown risks to the developing fetus. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with personalized neoantigen peptides and poly-ICLC, nursing women are excluded from this study.
* Individuals with history of an invasive malignancy are ineligible except for the following circumstances: a) individuals with a history of invasive malignancy are eligible if they have been disease -free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; b) individuals with the following cancers are eligible if diagnosed and treated: carcinoma in situ of the breast, oral cavity or cervix and basal cell or squamous cell carcinoma of the skin; c) individuals with prostate cancer managed with active surveillance that is not expected to limit their survival to <10 years.
* Participants with known CNS involvement
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to poly-ICLC.
* HIV-positive participants including those on combination antiretroviral therapy are ineligible because assessment of immunologic endpoints may be confounded by HIV-induced alterations in patient immune status and functio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2033-12-26 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Neovax following 4 weekly doses of rituximab assessed by the following | 2 years
  The proportion of all enrolled patients for whom sequencing and analysis leads to identification of at least 7 actionable peptides to initiate vaccine production and, of the patients who generate at least 7 actionable peptides, the proportion for whom the time from sample collection to vaccine availability is less than 12 weeks.

SECONDARY OUTCOMES:
The proportion of participants who achieve an IFN-γ T cell response to one or more of the peptide pools | 2 years
  The induction of IFN-γ T-cell response will be based on ELISPOT assessments taken prior to vaccine administration and at week 16 from both peripheral blood draws and bone marrow biopsies. The proportion of patients who achieve more than 55 SFU/106 PBMC or 3 times their baseline level will be presented with a 90% exact binomial confidence interval. Based on a cohort of size 10, the confidence interval will be no wider than 0.55. It is possible that the maximal response will occur at a different sampling time point or will vary between participants. Thus, this time point may vary from week 16.
The proportion of participants who convert from PR to CR | 2 years
  The investigators will report the proportion of patients converting from SD to CR/PR or from PR to CR based upon Lugano criteria in a descriptive fashion.
The proportion of participants who convert from SD to PR/CR | 2 years
  The investigators will report the proportion of patients converting from SD to CR/PR or from SD to PR or CR based upon Lugano criteria in a descriptive fashion.
Best Objective Response | 2 years
  The investigators will report the best objective response (CR, PR, SD, or PD) based upon Lugano criteria in a descriptive fashion.
To describe the safety and tolerability of NeoVax following 4 weekly doses of rituximab in patient with previously untreated follicular lymphoma | 2 years
  The investigators will report toxicity in a descriptive fashion using CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Reid W Merryman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No